CLINICAL TRIAL: NCT02338206
Title: Growth Hormone Adjuvant Therapy With Long Down Regulation Protocol in Poor Responders Undergoing In Vitro Fertilization Cycles: a Randomized Control Trial
Brief Title: Long Protocol and Growth Hormone in Poor Responders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, lecturer of obstetrics and gynecology, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP112015
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Infertility
Keywords: infertility
MeSH Terms: conditions — Infertility | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Long + Growth hormone (Active Comparator): Patients in this group were given a long protocol of pituitary down-regulation with triptorelin (Decapeptyl; Ferring, Switzerland) starting on the day 21 of preceding cycle at a dose of 0.1 mg/day, subcutaneously along with Growth hormone (Norditropin, Novo nordisk) co-treatment daily in a dose of 2.5 mg S.C. till the day of hCG administration.. On the second day of menstruation, Human menopausal gonadotrophin HMG (75 IU, Merional, IBSA) was started, and this was associated with reduction of triptorelin dose to 0.05 mg/day. This reduced daily dose, in addition to HMG and growth hormone, were continued till the day of hCG administration.
  Interventions: Drug: Growth hormone
- Long protocol only (No Intervention): Patients in this group were given a long protocol of pituitary down-regulation with triptorelin (Decapeptyl; Ferring, Switzerland) starting on the day 21 of preceding cycle at a dose of 0.1 mg/day, subcutaneously. On the second day of menstruation, Human menopausal gonadotrophin HMG (75 IU, Merional, IBSA) was started, and this was associated with reduction of triptorelin dose to 0.05 mg/day. This reduced daily dose, in addition to HMG, were continued till the day of hCG administration.

INTERVENTIONS:
Drug: Growth hormone
  Other Names: Norditropin, Novo nordisk
  Arms: Long + Growth hormone

SUMMARY:
The long down regulation protocol is widely used in the in vitro fertilization cycles, now it will be assessed regarding its efficacy, in poor responder females undergoing in vitro fertilization cycles, alone and after the addition of growth hormone.

ELIGIBILITY:
Inclusion Criteria:

* Poor responder females are those who posses two out of these three criteria:
* Female age ≥40 years
* Females who have at least one previous cancelled IVF cycle
* POR according to AFC ≤ 5 or low AMH value.

Exclusion Criteria:

* Females over 45 years
* Females with FSH more than 20 IU/l
* Females with previous ovarian surgery
* Females suffering from causes of infertility other than poor ovarian response
* Females refusing to be enrolled in the study

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Live birth rate | 12 months
  Fresh, Frozen, Cumulative

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Egypt

REFERENCES:
- [Derived] Dakhly DMR, Bassiouny YA, Bayoumi YA, Hassan MA, Gouda HM, Hassan AA. The addition of growth hormone adjuvant therapy to the long down regulation protocol in poor responders undergoing in vitro fertilization: Randomized control trial. Eur J Obstet Gynecol Reprod Biol. 2018 Sep;228:161-165. doi: 10.1016/j.ejogrb.2018.06.035. Epub 2018 Jun 22. PMID 29957401